CLINICAL TRIAL: NCT03216473
Title: A Multicenter, Double-blind, Randomized, Parallel, Active-controlled, Phase III Study to Evaluate the Efficacy and Safety of NEURONOX® vs. BOTOX® in Patients With Essential Blepharospasm
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Neuronox and Botox With Essential Blepharospasm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG1221MED
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Essential Blepharospasm
MeSH Terms: conditions — Benign essential blepharospasm | interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuronox (Experimental): Botulinum Toxin Type A for injection
  Interventions: Drug: Neuronox
- Botox (Active Comparator): Botulinum Toxin Type A for injection
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Neuronox — Clostridium Botulinum Toxin A 100 U
  Other Names: Botulinum Toxin Type A for injection
  Arms: Neuronox
Drug: Botox — Clostridium Botulinum Toxin A 100 U
  Other Names: Botulinum Toxin Type A for injection
  Arms: Botox

SUMMARY:
This clinical study evaluates the efficacy and safety of Neuronox compared with Botox in adults with essential blepharospasm.

DETAILED DESCRIPTION:
Subjects are randomly assigned into the two groups at the ratio of 1:1. The purpose of study is to confirm the non-inferiority of Neuronox to Botox in terms of the efficacy and safety in subjects with essential blepharospasm.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75
* Subjects had to have a confirmed clinical diagnosis of essential blepharospasm requiring treatment by injection

Exclusion Criteria:

* Subjects who underwent surgical operation
* Subjects with Neuroleptic induced blepharospasm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
JRS (Jankovic Rating Scale) sum-score | From baseline at 4 week
  Change from baseline at 4 week for the JRS (Jankovic Rating Scale) sum-score

IPD SHARING:
Plan to Share IPD: Undecided